CLINICAL TRIAL: NCT05622838
Title: Maternal alpha1 Antitrypsin as a Marker of Intrauterine Growth Restriction in Pre-eclamptic Women
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maryam Elwany Eldreemy, principal investigator, Assiut University
Other Study IDs: alpha1 antitrypsin as a marker
Record Dates: First submitted 2022-11-04; First posted 2022-11-21 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: alpha1 Anti-trypsin; Pre-Eclampsia; Intrauterine Growth Restriction
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Pre-Eclampsia; Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Pregnant Pre-eclamptic women with IUGR at 32-36 weeks
  Interventions: Diagnostic Test: Alpha1 -Antitrypsin level
- Pregnant Pre-eclamptic women with healthy fetus at 32-36 weeks
  Interventions: Diagnostic Test: Alpha1 -Antitrypsin level
- Normal pregnant women with healthy fetus
  Interventions: Diagnostic Test: Alpha1 -Antitrypsin level

INTERVENTIONS:
Diagnostic Test: Alpha1 -Antitrypsin level — measuring alpha1 -antitrypsin level in pregnant women

SUMMARY:
Intrauterine growth restriction (IUGR) is defined as a velocity of fetal growth less than the normal fetus growth potential for a specific neonate as per the race and gender. These neonates face many acute problems during peripartum and after birth .The causes of IUGR may be maternal, placental, fetal or genetic and also due to combination of any of these factors. Knowledge of etiologies of fetal growth restriction (FGR) is essential, so that future care can be targeted at prevention . It is apparent that FGR is primarily caused by placental dysfunction (PIH&PE), insufficiency that lead to reduced fetal growth overall. FGR is associated with lifelong burden of chronic diseases including metabolic, respiratory, cardiovascular and neurological deficits. Pre-eclampsia (PE) is diagnosed by the combined presentation of high blood pressure and proteinuria. New definitions also include maternal organ dysfunction, such as renal, liver, neurological or haematological complications, uteroplacental dysfunction, or FGR . In an attempt to correct fetus reduced supply the placenta release various cytokines and markers as Alpha-1 anti-trypsin (AAT). The Golgi apparatus secretes this cytokine in placental cytotrophoblast and blood vessels. AAT is antinflammatory antiprotease protective molecule. AAT rises during normal pregnancy. The suboptimal rise of AAT in pregnancy are liable for increased obstetrical complications like abortion, preterm labor. AAT levels were found decreased in placenta tissues from women with PE compared that of healthy women. Although AAT deficiency is associated with several pregnancy and placental disorders, little is known regarding AAT levels and PE .

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Pre-eclamptic women with IUGR at 32-36 weeks
* Pregnant Pre-eclamptic women with healthy fetus at 32-36 weeks
* Normal pregnant women with healthy fetus

Exclusion Criteria:

* Multiple pregnancy.
* Congenital fetal anomalies.
* Pregnant women with personal history of chronic hypertension.
* Pregnant women with renal failure.
* Pregnant women with cardiovascular disease.
* Pregnant women with diabetes mellitus.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Pregnant women with pre-eclampsia
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of serum alpha-1 anti-trypsin levels during pregnancy and their relationship with intrauterine growth restriction and pre eclampsia. | expected time of 2 years
  The levels of alpha-1 anti-trypsin will be measured in pregnant women and then will be correlated with the occurence of pre-eclampsia and intrauterine growth restriction

SECONDARY OUTCOMES:
Involvement of the results of this study in prediction and prevention of the disease. | expected time of 2 years
  The results that the investigators will get will be used as predictors and even preventers of intrauterine growth restriction which is a major problem threatening babies born to pre-eclamptic women

CONTACTS AND LOCATIONS:
Overall Officials: Omnia A Mohamed, Assistant professor, Study Chair — Clinical pathology department, Faculty of medicine, Assiut University, Egypt; Yousra M Mamdouh, Lecturer, Study Director — Clinical pathology department, Faculty of medicine, Assiut University, Egypt; Maryam E Eldreemy, Resident, Principal Investigator — Clinical pathology department, Faculty of medicine, Assiut University, Egypt

REFERENCES:
- [Background] Lee PA, Chernausek SD, Hokken-Koelega AC, Czernichow P; International Small for Gestational Age Advisory Board. International Small for Gestational Age Advisory Board consensus development conference statement: management of short children born small for gestational age, April 24-October 1, 2001. Pediatrics. 2003 Jun;111(6 Pt 1):1253-61. doi: 10.1542/peds.111.6.1253. PMID 12777538
- [Background] Hendrix N, Berghella V. Non-placental causes of intrauterine growth restriction. Semin Perinatol. 2008 Jun;32(3):161-5. doi: 10.1053/j.semperi.2008.02.004. PMID 18482615
- [Background] Bendix I, Miller SL, Winterhager E. Editorial: Causes and Consequences of Intrauterine Growth Restriction. Front Endocrinol (Lausanne). 2020 Apr 15;11:205. doi: 10.3389/fendo.2020.00205. eCollection 2020. No abstract available. PMID 32351451
- [Background] Mol BWJ, Roberts CT, Thangaratinam S, Magee LA, de Groot CJM, Hofmeyr GJ. Pre-eclampsia. Lancet. 2016 Mar 5;387(10022):999-1011. doi: 10.1016/S0140-6736(15)00070-7. Epub 2015 Sep 2. PMID 26342729
- [Background] Nori W, Ali AI. Maternal alpha-1-antitrypsin as a noval marker for growth restriction in pre-eclampsia. J Obstet Gynaecol Res. 2021 Dec;47(12):4250-4255. doi: 10.1111/jog.15043. Epub 2021 Sep 27. PMID 34571571